CLINICAL TRIAL: NCT01988974
Title: Feasibility Testing of the Alert for Atrial Fibrillation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Pamela J. McCabe, R.N., Ph.D., Assistant Professor of Nursing, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-007768
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alert for AF Program (Experimental): 1) participation in the Alert for Atrial Fibrillation program ) .
  Interventions: Behavioral: Alert for Atrial Fibrillation Program
- Attention control condition (Active Comparator): 2) participation in the healthy sleep program
  Interventions: Behavioral: Healthy Sleep

INTERVENTIONS:
Behavioral: Alert for Atrial Fibrillation Program — Participants' baseline knowledge of AF symptoms, and attitudes and beliefs about AF will be assessed using the KABAFS, and patients will receive cognitive-behavioral training directed toward survey responses associated with delay of treatment. Training will incorporate the content developed by the American College of Cardiology Foundation (ACCF), and participants will receive education about how to recognize an irregular pulse, and how to record the pulse rhythm in a daily log. The PI/RN coordinator will review the completed KABAFS to assess knowledge deficits, and identify attitudes and beliefs about AF that may hinder early treatment-seeking.
  Arms: Alert for AF Program
Behavioral: Healthy Sleep — Participants will receive a 45 minute face to face instruction about sleep hygiene
  Arms: Attention control condition

SUMMARY:
The purpose of this study is to determine the psychometric properties of the Knowledge, Attitudes, and Beliefs about Atrial Fibrillation Survey (KABAFS) and to generate critical, practical knowledge about the feasibility of conducting a randomized trial to test the effect of the Alert for Atrial Fibrillation program on treatment-seeking for symptoms of Atrial Fibrillation (AF).

DETAILED DESCRIPTION:
The purpose of the proposed research is to evaluate the psychometric properties of the Knowledge, Attitudes, and Beliefs about Atrial Fibrillation Survey (KABAFS), which is an instrument designed to tailor the delivery of the Alert for Atrial Fibrillation program. The proposed research will also test the feasibility of studying the effect of the Alert for Atrial Fibrillation program on treatment-seeking for symptoms of AF in a larger, randomized trial. This research is significant, because current research suggests that treatment seeking for AF is hindered when people do not recognize symptoms that represent AF, attribute those symptoms to alternative causes, or do not believe symptoms are serious enough to require medical evaluation. Interventions tailored to modify patient-specific knowledge, attitudes, and beliefs that hinder early treatment-seeking are critically needed in order to improve early detection of AF. The long term goal of this research is to improve health outcomes of those at risk for developing AF.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Under the care of providers from the Department of Medicine
* English-speaking
* Community dwelling,
* Have access to and ability to communicate via a telephone
* Have one or more risks for developing AF
* Not be diagnosed with AF

Exclusion Criteria:

* Documented cognitive impairment
* Uncompensated hearing or visual deficits
* Scheduled for surgery or have undergone a surgical procedure in the last 30 days,
* Undergoing active treatment for a malignancy
* Receiving hospice care will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes on the Knowledge, Attitudes, and Beliefs about Atrial Fibrillation Survey | Baseline, One Month, Two Months
  The KABAFS assesses patient knowledge of Atrial Fibrillation (AF) and the belief factors associated with delay in seeking treatment for AF. Participants will be measured at baseline (before the intervention), and then at 1 and 2 months after the intervention to identify if participants' knowledge and beliefs about treatment seeking have improved and continue to be improved from baseline as indicated by the KABAFS score.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J McCabe, PhD, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No